CLINICAL TRIAL: NCT05826509
Title: SUrGery With or Without dARolutamide in High-risk and/or Locally Advanced Prostate Cancer
Acronym: SUGAR
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22GENH03
Record Dates: First submitted 2023-04-12; First posted 2023-04-24 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Hight risk; Locally advanced; Radical prostatectomy; ADT sparing; Darolutamide
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (Active Comparator)
  Interventions: Other: Surgery alone
- Experimental arm (Experimental)
  Interventions: Drug: Peri-operative darolutamide + surgery.

INTERVENTIONS:
Other: Surgery alone — Radical prostatectomy with lymph node dissection will be performed.
  Arms: Control arm
Drug: Peri-operative darolutamide + surgery. — Darolutamide: 600 mg (2 tablets of 300 mg) twice daily with food, equivalent to a total daily dose of 1200 mg; for a total duration of 9 months. Darolutamide will start at day 1.
  Surgery: radical prostatectomy with lymph node dissection will be performed after at least 3 months of darolutamide treatment.
  Arms: Experimental arm

SUMMARY:
This is a phase II, multicenter, randomized open-label and comparative trial designed to study the effectiveness and the safety of androgen receptor antagonist (darolutamide) combined with surgery in patients with high-risk and/or locally advanced prostate cancer.

In this trial, patients will be assigned in one of the two following treatments arms:

* Arm A (control arm): Surgery alone (radical prostatectomy with lymph node dissection)
* Arm B (experimental arm): Peri-operative darolutamide + surgery (radical prostatectomy with lymph node dissection)

A total of 240 patients will have to be randomized with 120 patients in the control arm and 120 patients in the experimental arm.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Histologically confirmed adenocarcinoma of the prostate
3. High-risk and/or locally advanced prostate cancer diagnosis defined by:

   One of the following criteria is sufficient to define a high-risk and/or locally advanced prostate cancer:
   * ISUP grade 4 or 5 on biopsies
   * cN1 disease in MRI or PET-Scan
   * T3b disease in MRI

   If these criteria are not being identified, two of the following criteria are necessary to define high-risk and/or locally advanced prostate cancer:
   * PSA value >20 ng/ml
   * ≥ 50% of the core of biopsies need to be positive for adenocarcinoma ISUP grade 3
   * T3a disease in MRI
4. No distant metastasis confirmed by imaging (i.e., MRI/CT-Scan and Bone Scintigraphy or PET-Scan)
5. Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0-1
6. Patient eligible for radical prostatectomy as per the investigator
7. Adequate organ function within 28 days prior to start of treatment determined by the following central laboratory values:

   * Aspartate aminotransferase (AST), alanine aminotransferase (ALT), and total bilirubin less than the upper limit of normal (ULN; note that in subjects with Gilbert's syndrome, if total bilirubin is >1.5 X ULN, measure direct and indirect bilirubin. If direct bilirubin is ≤1.5 X ULN, the subject may be eligible);
   * Serum creatinine <1.5 mg/dL;
   * Platelets ≥75,000/uL, without transfusion and/or growth factors within 1 month prior to randomization;
   * Hemoglobin >12.0 g/dL (7.4 mmol), without transfusion and/or growth factors within 1 month prior to randomization;
   * Adequate renal function: creatinine clearance/eGFR within normal limits to baseline assessed as per local standard method;
   * Normal cardiac function according to local standard by 12-lead Electrocardiogram (ECG) (complete, standardized 12-lead recording).
8. Patient able to receive darolutamide for up to 9 months as per the investigator
9. Patient able to swallow whole study drug tablets
10. Life expectancy more than 5 years
11. Men engaged in sexual activity with a woman of childbearing potential should accept (or female partners of men enrolled in the study who are of childbearing potential or are pregnant) to use an highly effective contraception during darolutamide treatment and at least one week after the end of the investigational product
12. Signed informed consent
13. Patient able to participate and willing to give informed consent prior performance of any study-related procedures and to comply with the study protocol for the duration of the study, including undergoing treatment and scheduled visits and examinations including follow up
14. Patient affiliated to a Social Health Insurance in France.

Exclusion Criteria:

1. Distant metastasis (clinical stage M1). Nodal disease below the iliac bifurcation (clinical stage N1) is not an exclusion.
2. Pathological finding consistent with small cell, ductal or neuroendocrine carcinoma of the prostate
3. Prior treatment for prostate cancer
4. Castrated men (Bilateral orchiectomy or other)
5. History of any pelvic radiation
6. Any of the following concurrent illness within 6 months prior to first dose of study drug: severe or unstable angina, myocardial infarction, symptomatic congestive heart failure, arterial or venous thromboembolic events (eg, pulmonary embolism, cerebrovascular accident including transient ischemic attacks), or clinically significant ventricular arrhythmias or New York Heart Association Class II to IV heart disease; uncomplicated deep vein thrombosis is not considered exclusionary
7. Uncontrolled hypertension as indicated by a systolic blood pressure (BP) ≥ 160 mmHg or diastolic BP ≥ 100 mmHg at screening despite medical management. Participants with hypertension can enroll provided BP is stable and controlled by anti-hypertensive treatment
8. HIV-positive patient with one or more of the following: Not receiving highly active antiretroviral therapy; Had a change in antiretroviral therapy within 6 months of the start of screening; Receiving antiretroviral therapy that may interfere with study drug; CD4 count <350 at screening; AIDS-defining opportunistic infection within 6 months of start of screening
9. Active or symptomatic viral hepatitis or chronic liver disease; ascites or bleeding disorders secondary to hepatic dysfunction
10. Gastrointestinal conditions affecting absorption
11. Known or suspected contraindications or hypersensitivity to darolutamide
12. Treatment with strong CYP3A4 inducers and P-gp inducers within 2 weeks or 5 drug-elimination half-lives, whichever is longer, prior to initiation of study drug
13. Major surgery within 28 days before first dose of study treatment
14. Any psychological, familial, geographic or social situation, according to the judgment of investigator, potentially preventing the provision of informed consent or compliance to study procedure
15. Patient who has forfeited his/her freedom by administrative or legal award or who is under legal protection (curatorship and guardianship, protection of justice)
16. Concurrent enrolment in another interventional therapeutic clinical study.
17. Patients with a history of another malignancy at high risk of recurrence within 5 years and with a concurrent malignancy requiring active treatment or having required anticancer treatment within 6 months prior to inclusion.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-08-10 (Actual); Primary Completion 2031-02 (Estimated); Study Completion 2031-02 (Estimated)

PRIMARY OUTCOMES:
The non-curable progression-free survival (NC-PFS) defined as the time from randomization to non-curable event. | 5 years for each patient

SECONDARY OUTCOMES:
Metastatic-Free Survival (MFS) defined as the time from randomization to the appearance of distant metastasis or death from any cause. | 5 years for each patient
PSA-RFS (Recurrence-Free survival) defined as the time from randomization to PSA recurrence according to the European Association of Urology (EAU) criteria or death from any cause. | 5 years for each patient
Overall Survival (OS) defined as the time from randomization to death from any cause. | 5 years for each patient
pathological Complete Response (pCR) rate defined as the number of patients presenting a pathological complete response (i.e., absence of residual tumor found in the surgery specimens) divided by the number of patients in the experimental arm. | 5 years for each patient
Safety assessed using the NCI-CTCAE Version 5.0. | 3 years for each patient
Quality of life will evaluated using the Functional Assessment of Cancer Therapy-Prostate (FACT-P) questionnaire. | 1 year for each patient
  Subscale Domains: Physical Well-Being, Social/Family Well-Being, Emotional Well-Being, Functional Well-Being, Prostate Cancer Subscale.
  Responses to questions use a five-point Likert-type scale ranging from 0 ("not at all") to 4 ("very much so").
Quality of life will evaluated using the 5-level EuroQol 5-Dimensional (EQ5D-5L) questionnaire. | 1 year for each patient
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems.
Quality of life will evaluated using the International Prostate Symptom Score (IPSS) questionnaire. | 1 year for each patient
  The I-PSS is based on the answers to seven questions concerning urinary symptoms. Each question is assigned points from 0 (never) to 5 (almost always).
Quality of life will evaluated using the International Index of Erectile Function (IIEF-15) questionnaire. | 1 year for each patient
  The IIEF is a 15-item questionnaire containing five domains including erectile function, orgasmic function, sexual desire, intercourse satisfaction, and overall satisfaction. Each item is rated from 0 (or 1) (Severe ED/No sexual activity) to 5 (Mild/No ED).

CONTACTS AND LOCATIONS:
Locations (20):
- France (20):
  - Chu Angers, Angers
  - CHU Bordeaux, Bordeaux
  - Institut Bergonié, Bordeaux
  - Chu Henri Mondor, Créteil
  - CHU Grenoble, Grenoble
  - Hopital Claude Huriez, Lille
  - CHU Lyon - Hôpital Edouard Herriot, Lyon
  - Institut Paoli-Calmettes, Marseille
  - Hopital Paris Saint-Joseph, Paris
  - Hopital Bichat - Ap-Hp, Paris
  - Hopital Europeen Georges-Pompidou, Paris
  - Hopital Pitie Salpetriere, Paris
  - Institut Mutualiste Montsouris, Paris
  - CHU Lyon - Sud, Pierre-Bénite
  - Clinique La Croix Du Sud, Quint-Fonsegrives
  - CHU Rennes, Rennes
  - Hopital Foch, Suresnes
  - CHU Toulouse, Toulouse
  - Institut Universitaire Du Cancer Toulouse - Oncopole, Toulouse
  - Chu Tours - Hopital Bretonneau, Tours